CLINICAL TRIAL: NCT06002542
Title: Mobile Chat Service for Parents of Children in Pediatric Emergency Room: A Randomized Control Study
Brief Title: Mobile Chat Service for Parents of Children in Pediatric Emergency Room
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TMI
Record Dates: First submitted 2023-08-01; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Medical Informatics; Pediatric Emergency Medicine; Emergency Medicine

STUDY DESIGN:
Intervention Model Description: open-label randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information provided (Experimental): Participants are invited to the chat room and receive messages, which include the stages of their medical care, information about tests and medications, and non-medical information such as directions to pharmacy and parking information.
  Interventions: Behavioral: Information provided
- Control (Experimental): Participants are invited to the chat room and they can get information when they request it.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Information provided — get information at every stage of care in emergency room
  Arms: Information provided
Behavioral: Control — Information is only provided when participants request it.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to test giving all medical/non-medical information in the pediatric emergency room(ER).

Main questions it aims to answer are:

* Does providing medical/non-medical information to parents of patients visiting the emergency room raise the satisfaction with the ER visit?
* Does providing medical/non-medical information to parents of patients visiting the emergency room lower the workload of medical staff?

  60 participants will be randomly assigned to treatment group and control group. Both groups will communicate freely with the researchers through mobile chat service. Treatment group will get information of medical/non-medical information in emergency room and control group will get information if they need. Before leaving the emergency room, both group will fill out a questionnaire related to satisfaction with the emergency room visits. 5 out of 30 participants of each group will be interviewed about their satisfaction with service.

  10 nurses in charge of patients participating in the study record the number of questions directly received and 5 out of 10 nurse will be interviewed about their nursing experience for participants using mobile chatbot service.

Researchers will compare treatment group and control group to see if providing medical/non-medical information raise the satisfaction with emergency room visits.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test giving all medical/non-medical information in the pediatric emergency room.

Main questions it aims to answer are:

* Does providing medical/non-medical information to parents of patients visiting the emergency room raise the satisfaction with the ER visit?
* Does providing medical/non-medical information to parents of patients visiting the emergency room lower the workload of medical staff?

Design :

60 participants will be randomly assigned to treatment group and control group. Both groups will communicate freely with the researchers through mobile chat service. Treatment group will get information of medical/non-medical information in emergency room and control group will get information if they need. Before leaving the emergency room, both group will fill out a questionnaire related to satisfaction with the emergency room visits.

5 out of 30 participants of each group will be interviewed about their satisfaction with service.

10 nurses in charge of patients participating in the study record the number of questions directly received and 5 out of 10 nurse will be interviewed about their nursing experience for participants using mobile chatbot service.

Researchers will compare treatment group and control group to see if providing medical/non-medical information raise the satisfaction with emergency room visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Parents of patients whose KTAS(Korean Triage and Acuity Scale) is 2, 3, 4.
* Parents of patients whose chief complaints are fever, abdominal pain, dyspnea, nausea and vomiting, and skin rash.
* Those who voluntarily agreed to participate in the study.

Exclusion Criteria:

* Those who didn't consent to participate in the study.
* Parents of patients whose KTAS(Korean Triage and Acuity Scale) is 1 or 5.
* Those who doesn't use mobile phone or those who don't have the appropriate level of consciousness to send and receive messages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
ED CAHPS(Emergency department Consumer Assessment of Healthcare Providers and System) Questionnaire score at discharge | Discharge time, 6 hours on average from arriving emergency room.
  ED CAHPS is a survey instrument for measuring patients' experience of care in emergency department.

SECONDARY OUTCOMES:
Interview for participants | After leaving the emergency room visit, within 48hours
  Interview on the experience and satisfaction of using mobile chatbot services

OTHER OUTCOMES:
Questions to nurse | average of 6 hours from the time participants arrived at the emergency room to discharge.
  The nurse in charge counts the number of questions received from participants.
Interview for nurse | After work, within 48hours after nursing participants.
  Interviewing whether chatbot services lower their tasks

CONTACTS AND LOCATIONS:
Overall Officials: Wonchul Cha, PhD, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ED CAHPS survey and guideline — https://www.cms.gov/Research-Statistics-Data-and-Systems/Research/CAHPS/ED